CLINICAL TRIAL: NCT00599352
Title: Hypovitaminosis D and an Inadequate PTH Response in Chronic Liver Disease Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Rajib Bhattacharya, MD (Other)
Responsible Party: Sponsor-Investigator, Rajib Bhattacharya, MD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11152; CRA # 10345
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Liver Disease; Hypovitaminosis
Keywords: Hypovitaminosis; Chronic liver disease
MeSH Terms: conditions — Avitaminosis | interventions — Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Magnesium infusion
  Interventions: Dietary Supplement: magnesium

INTERVENTIONS:
Dietary Supplement: magnesium — Single infusion of elemental magnesium given over 4 hours, 0.2mEq/kg (2.4 mg/kg)

SUMMARY:
The purpose of this study is to determine how common low levels of magnesium are in patients with end stage liver disease. In addition, investigator is trying to determine if low levels of magnesium affect the release of parathyroid hormone in patients with end stage liver disease and low vitamin D levels

DETAILED DESCRIPTION:
Hypovitaminosis D is a common condition found in patients referred for orthotopic liver transplant. The classical physiologic response to vitamin D deficiency is the development of secondary hyperparathyroidism. However, several previous studies have found a high incidence of inappropriate functional hypoparathyroidism in patients with chronic liver disease and hypovitaminosis D. The mechanism underlying this functional hypoparathyroidism is not understood but previous investigators have postulated that it is related to intracellular magnesium (Mg) deficiency. Our short term goals of this pilot project are two fold: (a) We will estimate the prevalence of magnesium deficiency in chronic liver disease patients by performing standard Mg loading testing (b) We will examine the effects of acute intravenous Mg infusion on the calcium-PTH axis. The vitamin D-PTH endocrine system is one of the principal regulators of calcium homeostasis and bone metabolism. Metabolic bone disease is a quite pervasive problem in chronic liver disease patients. Insight into this important endocrine system will aid us in our long term goals of addressing metabolic bone disease issues in this patient population.

ELIGIBILITY:
Inclusion Criteria:

chronic liver disease patients > 18 years of age Diagnosed end stage liver disease >18 years of age Presence of hypovitaminosis D Glomerular filtration rate of 60 ml/min./1.73m2 or greater

Exclusion Criteria:

subjects with known parathyroid disease subjects taking magnesium supplementation <18 years of age History of parathyroid disease Current supplementation of magnesium Abnormal baseline EKG Current diagnosis of cancer or undergoing cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Perform a standard magnesium loading test to determine urinary magnesium retention in order to define prevalence of magnesium insufficiency in a chronic liver disease population | One Month

SECONDARY OUTCOMES:
Evaluate the effects of intravenous magnesium loading on the calcium-PTH endocrine axis by measuring pre and immediate post infusion calcium and PTH | One Month

CONTACTS AND LOCATIONS:
Overall Officials: Rajib Bhattacharya, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States